CLINICAL TRIAL: NCT05374733
Title: Coronary Physiology Peri-Transcatheter Left-sided Valvular Interventions in Patients With Severe Aortic Stenosis or Mitral Regurgitation
Brief Title: Coronary Physiology Peri-Transcatheter Left-sided Valvular Interventions
Acronym: POTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Prof. Dr. Nicolas M. Van Mieghem, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POTUS
Record Dates: First submitted 2021-09-21; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Aortic Valve Stenosis; Mitral Regurgitation; Coronary Artery Disease; Fractional Flow Reserve
Keywords: Coronary Physiology
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, observational study with invasive measurements in two cohorts (TAVI cohort and TMVr cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm (Other): Coronary physiology measurements both pre- and post- transcatheter left-sided valvular intervention.
  Interventions: Diagnostic Test: Coronary Physiology assessment

INTERVENTIONS:
Diagnostic Test: Coronary Physiology assessment — 1. Pd/Pa, diastolic pressure ratio (dPR), resting full cycle ratio (RFR), FFR, coronary flow reserve (CFR), and index of microvascular resistance (IMR) measurements in the coronary of interest before the valvular intervention.
  2. Pd/Pa, dPR, RFR, FFR, vFFR, CFR and IMR measurements in the coronary of interest after the valvular intervention.

SUMMARY:
Prospective, single-arm, observational study with invasive coronary physiology measurements before and after transcatheter left-sided valvular intervention.

DETAILED DESCRIPTION:
The POTUS study is a prospective, investigator-initiated, single-arm observational study with invasive measurements that will consist of two cohorts. The first cohort consists of 120 patients with intermediate coronary artery disease who undergo a transcatheter aortic valve implantation (TAVI) for severe aortic valve stenosis ('TAVI cohort'). The second cohort consists of 30 patients with intermediate coronary artery disease who undergo transcatheter mitral valve repair (TMVr) for functional/degenerative mitral regurgitation ('TMVr cohort'). Both cohorts will undergo a battery of coronary physiological tests both before and after the valvular intervention. Additionally, in the case that the fractional flow reserve (FFR) over a coronary lesion is significant (i.e. FFR ≤ 0.80) during the post valvular intervention measurements, additional percutaneous coronary intervention (PCI) will take place during the same procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* a) TAVI cohort: severe aortic valve stenosis for which TAVI is scheduled after discussion in the Heart Team.

  b) TMVr cohort: severe functional/degenerative mitral regurgitation for which TMVr is scheduled after discussion in the Heart Team.
* At least intermediate coronary artery disease, defined as 50-99% diameter stenosis in a vessel ≥ 2.5 mm
* Elective procedure
* Written informed consent

Exclusion Criteria:

* TAVI cohort: height coronary ostia < 10 mm
* Severe chronic kidney disease, defined as estimated glomerular filtration rate < 30 ml/min.
* Contra-indication for intravenous adenosine: severe asthma or chronic obstructive pulmonary disease, known allergy to adenosine or previous reported bronchospasm in response to adenosine.
* Degenerated surgical or transcatheter aortic valve bioprosthesis.
* Vessels that have collaterals to a chronic total occlusion or that are supplied by an arterial or venous bypass graft will not be interrogated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The change in the FFR value before and after TAVI | Directly before and after the TAVI procedure (1 hour)
  The impact of TAVI on FFR
The change in the FFR value before and after TMVr | Directly before and after the TMVr procedure (1 hour)
  The impact of TMVr on FFR

SECONDARY OUTCOMES:
The change in RFR before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on RFR
The change in dPR before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on dPR
The change in Pd/Pa before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on Pd/Pa
The change in CFR before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on CFR
The change in IMR before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on IMR
The change in transvalvular gradient before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on the transvalvular gradient
The change in left ventricular end-diastolic pressure (LVEDP) before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on the LVEDP
The change in systemic aortic pressure before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on hemodynamics
The change in heart rate before and after transcatheter valvular intervention (either TAVI or TMVr) | Directly before and after the TAVI/TMVr procedure (1 hour)
  The impact of TAVI/TMVr on hemodynamics

OTHER OUTCOMES:
The difference in the mean change in the FFR between the TAVI cohort and the TMVR cohort. | Baseline
  The mean change in the FFR in TAVI patients will be compared to mean change in FFR in TMVr patients.
The difference in the mean change in the RFR between the TAVI cohort and the TMVR cohort. | Baseline
  The mean change in the RFR in TAVI patients will be compared to mean change in RFR in TMVr patients.
The difference in the mean change in the dPR between the TAVI cohort and the TMVR cohort. | Baseline
  The mean change in the dPR in TAVI patients will be compared to mean change in dPR in TMVr patients.
The difference in the mean change in the Pd/Pa between the TAVI cohort and the TMVR cohort. | Baseline
  The mean change in the Pd/Pa in TAVI patients will be compared to mean change in Pd/Pa in TMVr patients.
The number of patients in who the post FFR, RFR, Pd/Pa or dPR value crosses the border of hemodynamic significance as compared to the value pre-valvular intervention. | Baseline
  Number of patients who have 1) a positive FFR/RFR/Pd/Pa/dPR value pre-valvular intervention, and negative FFR/RFR/Pd/Pa/dPR post-valvular intervention or 2) a negative FFR/RFR/Pd/Pa/dPR pre-valvular intervention, and positive FFR/RFR/Pd/Pa/dPR value post-valvular intervention.
The number of patients in whom the decision for coronary revascularization is altered when based on the post-procedural FFR value instead of angiographic stenosis severity. | Baseline
  Number of patients who have 1) post-valvular intervention FFR ≤ 0.80 and diameter stenosis 50-70% or 2) post-valvular intervention FFR > 0.80 and diameter stenosis ≥ 70%.
The diagnostic performance of vessel FFR (vFFR; an angiography-based FFR index) in the setting of valvular heart disease. | Baseline
  The vFFR pre-intervention will be validated against the FFR-value both pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No